CLINICAL TRIAL: NCT02071979
Title: Effectiveness of Autologous Platelet Rich Plasma in the Treatment of Chronic Skin Wounds
Brief Title: Registry Trial of the Effectiveness of Platelet Rich Plasma for Chronic Non-Healing Wounds
Acronym: CMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Arteriocyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ART-13-006; CAG-00190R3 (Other: CMS)
Record Dates: First submitted 2014-02-20; First posted 2014-02-26 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Diabetic Foot Ulcers; Venous Ulcers; Pressure Ulcers
Keywords: Chronic; Non-healing; Wounds
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Pressure Ulcer; Bronchiolitis Obliterans Syndrome; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Autologous PRP Gel (Experimental): The method of application for PRP treatment will be decided by the clinician in accordance with the appearance of the wound bed. The application of topical PRP gel may be used in chronic wounds possessing an open, moist wound bed according to following treatment schedule: Baseline/Week 0, Week 1, Week 2, Week 3, Week 7, and Week 11. The Arteriocyte Magellan® System (510(k) cleared) will be used to prepare the autologous PRP gel. For data analysis, the data from these patients will be classified as PRP Treatment Group (Topical application) data.
  Interventions: Device: Autologous PRP Gel; Procedure: Standard Wound Care
- Autologous PRP Injections (Experimental): The method of application for PRP treatment will be decided by the clinician in accordance with the appearance of the wound bed. Autologous PRP Injections may be used where chronic wounds possess a raised, hyperproliferative wound margin and/or plaque, according to following treatment schedule: Baseline/Week 0, Week 1, Week 2, Week 3, Week 7, and Week 11. The Arteriocyte Magellan® System (510(k) cleared) will be used to prepare Autologous PRP for injections. For data analysis, the data from these patients will be classified as PRP Treatment Group (Direct Injection) data.
  Interventions: Device: Autologous PRP Injections; Procedure: Standard Wound Care
- Autologous PRP Gel plus PRP Injections (Experimental): The method of application for PRP treatment will be decided by the clinician in accordance with the appearance of the wound bed. Some wounds may be suitable for both Autologous PRP Gel plus PRP Injections. Autologous PRP injections into, or to the periphery of, a moist wound bed in which no scarification or raised wound margin is apparent (where autologous PRP Gel can also be used) may further augment wound healing by addressing wound healing in multiple areas, following the treatment schedule: Baseline/Week 0, Week 1, Week 2, Week 3, Week 7, and Week 11. The Arteriocyte Magellan® System (510(k) cleared) will be used to prepare the autologous PRP gel. For data analysis, the data from these patients will be classified as PRP Treatment Group (Topical and Direct) data.
  Interventions: Device: Autologous PRP Gel; Device: Autologous PRP Injections; Device: Autologous PRP Gel plus PRP Injections; Procedure: Standard Wound Care
- Standard Wound Care (No Intervention): Subjects in the control group will receive Standard Wound Care treatment for chronic wounds according to accepted medical practices. For data analysis, the data from these patients will be classified as Control (Standard of Care) Group data

INTERVENTIONS:
Device: Autologous PRP Gel — Autologous PRP Gel is prepared using the Arteriocyte Magellan® System (510(k) approved), an Autologous Platelet Separator Instrument, which is a microprocessor-controlled centrifuge designed to be used in the clinical laboratory or intraoperatively at point of care for the safe and rapid preparation of platelet poor plasma and platelet concentrate (platelet rich plasma) from a small sample of blood. The Arteriocyte Magellan® automatically and quickly separates PRP from anticoagulated blood and dispenses it into a separate sterile syringe. The prepared PRP is then activated (by mixing with thrombin and calcium chloride) and sprayed directly on the area to be treated.
  Arms: Autologous PRP Gel; Autologous PRP Gel plus PRP Injections
Device: Autologous PRP Injections — Autologous PRP Gel is prepared using the Arteriocyte Magellan® System (510(k) approved), an Autologous Platelet Separator Instrument, which is a microprocessor-controlled centrifuge designed to be used in the clinical laboratory or intraoperatively at point of care for the safe and rapid preparation of platelet poor plasma and platelet concentrate (platelet rich plasma) from a small sample of blood. The Arteriocyte Magellan® automatically and quickly separates PRP from anticoagulated blood and dispenses it into a separate sterile syringe. The prepared PRP is then drawn into multiple small syringes and injected directly into the wound bed or the skin surrounding it.
  Arms: Autologous PRP Gel plus PRP Injections; Autologous PRP Injections
Device: Autologous PRP Gel plus PRP Injections — Autologous PRP Gel is prepared using the Arteriocyte Magellan® System (510(k) approved), an Autologous Platelet Separator Instrument, which is a microprocessor-controlled centrifuge designed to be used in the clinical laboratory or intraoperatively at point of care for the safe and rapid preparation of platelet poor plasma and PRP from a small sample of blood. The Arteriocyte Magellan® automatically and quickly separates PRP from anticoagulated blood and dispenses it into a separate sterile syringe. The prepared PRP is then divided into equal parts and half is drawn into multiple small syringes and injected directly into the skin surrounding the wound bed, half is activated (by mixing with thrombin and calcium chloride) and sprayed the wound bed.
  Arms: Autologous PRP Gel plus PRP Injections
Procedure: Standard Wound Care — Subjects in the control group will receive Standard Wound Care treatment for chronic wounds according to accepted medical practices.
  Arms: Autologous PRP Gel; Autologous PRP Gel plus PRP Injections; Autologous PRP Injections

SUMMARY:
This study will examine differences in the process of wound-healing in patients treated with platelet rich plasma (a concentration of proteins derived from a patients own blood) applied to the wound as a gel; injected into the wound or surrounding tissue; or both; compared to patients treated with usual medical treatment . This study seeks to enroll patients who are 18 or older with a non-healing skin wound that is at least 30 days old. Only patients with Diabetic Foot Ulcers, Venous Ulcers, or Pressure Ulcers will be included in the study.

DETAILED DESCRIPTION:
The proposed investigation is designed to solicit a large number of patients (N=1,500) with non-healing wounds (Diabetic Foot Ulcers, Venous Ulcers, or Pressure Ulcers) that have not responded to standard wound care in the previous 30 days or more. A prospective, interventional, single-blinded, controlled, registry trial will be used. Data will be analyzed to compare patients who received PRP therapy (PRP gel application, PRP injection, or both) and standard wound care (usual customary care) with patients who received standard wound care (usual customary care), only. Wound size, rate of healing, quality of life, and recurrence of wound will be measured during the 16-week period at usual office visits.

Hypotheses to be tested:

1. Treatment of a chronic wound with standard of care and autologous platelet rich plasma (PRP) will increase the velocity of healing (rate of wound closure) over a twenty week period as compared to patients receiving standard wound care only (Control Group), which results in the patient's ability to return to previous function and resumption of normal activities.
2. Treatment of a chronic wound with standard of care and autologous platelet rich plasma (PRP) will result in complete wound healing within twenty weeks, whereas complete wound healing will not be observed within twenty weeks in patients receiving standard wound care only (Control Group).

ELIGIBILITY:
Inclusion Criteria:

* Medicare Eligible
* Written informed consent obtained from either the subject or the subject's legally acceptable representative prior to screening activities
* Male or female ≥ 18 years of age
* Duration of Diabetic Foot Ulcers (DFU),Venous Ulcers (VU), or Pressure Ulcers (PU) is greater than 30 days at first visit/subject screening
* DFU is classified as Wagner 1 -2 on the Wagner classification system
* If more than one non-healing wound is present, the largest of the wounds that is classified as a Wagner 1 - 2.
* If a subject has multiple eligible wounds, the largest wound will be selected. There must be at least 4 cm between the index wound and other wounds; if all wounds are closer than 4 cm, the subject should not be enrolled (screen failure).
* The ulcer must be clinically non-infected
* Able and willing to comply with the procedures required by the protocol. Subjects may be managed as either inpatient or outpatient.
* If a female of childbearing potential, the subject must have a negative urine pregnancy test at screening and must agree to use adequate contraception methods for the duration of the study.
* Ankle Brachial Index (ABI) greater than or equal to 0.7.

Exclusion Criteria:

* Subjects with known sensitivity to components of the Arteriocyte BioBandage™ (calcium chloride, thrombin, acid citrate dextrose solution A (ACDA)).
* Current treatment of another chronic wound in the same limb (defined as arm or leg).
* Wound is not of DFU, PU, or VU pathophysiology.
* PU is classified as late stage III or stage IV.
* Confirmed presence of osteomyelitis, or if osteomyelitis is suspected.
* Received systemic corticosteroids or immunosuppressive agents, hyperbaric oxygen therapy (HBOT), electrostimulation, growth factors, or any cell or tissue-derived products for wounds during the 30 days preceding the screening visit.
* Any chronic condition requiring the use of systemic corticosteroids 30 days prior to study entry and anytime during the course of the study.
* Received radiation therapy or chemotherapy within previous 6 months.
* Any malignancy other than non-melanoma skin cancer.
* Patient has radiographic evidence consistent with diagnosis of neuropathic osteoarthropathy (Charcot foot) in the treatment limb.
* Ulcer area decreases by greater than or equal to 30% during screening period
* Subjects who are cognitively impaired and do not have a healthcare proxy.
* Subject has inadequate venous access for repeated blood draw required for PRP preparation.
* Subject has sickle cell anemia.
* Subject is pregnant or plans to become pregnant during the duration of the trial.
* Concurrent participation in a clinical trial in which an investigational agent is used.
* Females who are nursing.
* Subjects with Thrombocytopenia < 100,000 platelets/µL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Wound Size | 16 Weeks
  Wound size will be measured with ruler/probe for length, width and depth as well as with digital imaging. Wound size will be assessed in digital images taken of the wound.

SECONDARY OUTCOMES:
Rate of wound closure (change in wound size over time) | 16 weeks
  The ratio of wound percent change over time will be used
Complete wound healing | 16 weeks
  Complete wound healing is determined when the wound shows no sign of drainage for two consecutive visits (over two weeks)
Health Related Quality of Life | 16 weeks
  The Center for Disease Control (CDC) Health Related Quality of Life (HRQoL)-14, "Healthy Days Measure" will be administered
Wound recurrence | 16 weeks
  Incidence of wound recurrence over the course of 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Hamilton, Study Director — Compass Biomedical (Formerly Arteriocyte, Inc.)
Locations (6):
- United States (6):
  - Good Samaritan Wound Care Center, Bakersfield, California
  - Sunnyside Foot and Ankle, Idaho Falls, Idaho
  - Wound Care Center, Englewood Hospital and Medical Center, Englewood, New Jersey
  - Comprehensive Wound Healing Center and Hyperbarics, Lake Success, New York
  - Total Foot Care, Cleveland, Ohio
  - Heritage Valley Health System, Beaver, Pennsylvania

REFERENCES:
- [Background] Mustoe TA, O'Shaughnessy K, Kloeters O. Chronic wound pathogenesis and current treatment strategies: a unifying hypothesis. Plast Reconstr Surg. 2006 Jun;117(7 Suppl):35S-41S. doi: 10.1097/01.prs.0000225431.63010.1b. PMID 16799373
- [Background] Martinez-Zapata MJ, Marti-Carvajal AJ, Sola I, Exposito JA, Bolibar I, Rodriguez L, Garcia J. Autologous platelet-rich plasma for treating chronic wounds. Cochrane Database Syst Rev. 2012 Oct 17;10:CD006899. doi: 10.1002/14651858.CD006899.pub2. PMID 23076929
- [Background] Lacci KM, Dardik A. Platelet-rich plasma: support for its use in wound healing. Yale J Biol Med. 2010 Mar;83(1):1-9. PMID 20351977
- [Background] Crovetti G, Martinelli G, Issi M, Barone M, Guizzardi M, Campanati B, Moroni M, Carabelli A. Platelet gel for healing cutaneous chronic wounds. Transfus Apher Sci. 2004 Apr;30(2):145-51. doi: 10.1016/j.transci.2004.01.004. PMID 15062754
- [Background] Mazzucco L, Medici D, Serra M, Panizza R, Rivara G, Orecchia S, Libener R, Cattana E, Levis A, Betta PG, Borzini P. The use of autologous platelet gel to treat difficult-to-heal wounds: a pilot study. Transfusion. 2004 Jul;44(7):1013-8. doi: 10.1111/j.1537-2995.2004.03366.x. PMID 15225241
- [Background] Shan GQ, Zhang YN, Ma J, Li YH, Zuo DM, Qiu JL, Cheng B, Chen ZL. Evaluation of the effects of homologous platelet gel on healing lower extremity wounds in patients with diabetes. Int J Low Extrem Wounds. 2013 Mar;12(1):22-9. doi: 10.1177/1534734613477113. PMID 23509083
- [Background] Yang HS, Shin J, Bhang SH, Shin JY, Park J, Im GI, Kim CS, Kim BS. Enhanced skin wound healing by a sustained release of growth factors contained in platelet-rich plasma. Exp Mol Med. 2011 Nov 30;43(11):622-9. doi: 10.3858/emm.2011.43.11.070. PMID 21847007
- [Background] Driver VR, Hanft J, Fylling CP, Beriou JM; Autologel Diabetic Foot Ulcer Study Group. A prospective, randomized, controlled trial of autologous platelet-rich plasma gel for the treatment of diabetic foot ulcers. Ostomy Wound Manage. 2006 Jun;52(6):68-70, 72, 74 passim. PMID 16799184